CLINICAL TRIAL: NCT03765775
Title: A Randomized, Phase II Study of Anlotinib Combined With Sintilimab(IBI 308) in First-generation EGFR-TKIs Drug Resistance Along With T790M Negative NSCLC
Brief Title: Anlotinib Plus Sintilimab for NSCLC Patients With First-generation EGFR-TKIs Drug Resistance Along With T790M Negative
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Hospital of Shijiazhuang City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC01
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma; Non-small Cell Lung Cancer; Lung Neoplasm
Keywords: Non-small Cell Lung Cancer; Anlotinib; Sintilimab
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — sintilimab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride+Sintilimab (Experimental): Participants receive Sintilimab (IBI 308) 200 mg, administered as intravenous (IV) infusion on Day 1 of each 21-day cycle , Anlotinib 12mg, administered as PO on Day1-14 of each 21-day cycle until documented PD
  Interventions: Biological: Sintilimab; Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Biological: Sintilimab — Participants receive Sintilimab(IBI 308) 200 mg, administered as intravenous (IV) infusion on Day 1 of each 21-day cycle
Drug: Anlotinib Hydrochloride — Participants receive Anlotinib 10 mg, administered as PO on Day 1-14 of each 21-day cycle
  Other Names: Anlotinib

SUMMARY:
This is an efficacy and safety study of Anlotinib combined with Sintilimab (IBI 308) in participants with advanced or metastatic non-small cell lung cancer (NSCLC) who have received first-generation EGFR-TKIs resistance along with T790M negative.

DETAILED DESCRIPTION:
Participants receive Sintilimab(IBI 308) 200 mg, administered as intravenous (IV) infusion on Day 1, Anlotinib 12mg, administered as PO on Day1-14 of each 21-day cycle until documented PD.The primary hypothesis of this study is that participants will have a longer Progression Free Survival (PFS), as assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) when treated with Anlotinib plus Sintilimab(IBI 308).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects volunteered to participate in this study and signed the informed consent form, with good compliance and follow-up.
2. Male or female patients aged 18-75 years old.
3. Has a histologically-confirmed or cytologically confirmed diagnosis of stage IV nonsquamous NSCLC.

   Has confirmation that epidermal growth factor receptor (EGFR) mutation，with first-generation EGFR-TKIs drug resistance T790M negative .
4. Has measurable disease.
5. There is at least one target lesion that has not received radiotherapy in the past 3 months, and it can be accurately measured in at least one direction (the maximum diameter needs to be recorded) by magnetic resonance imaging (MRI) or computed tomography (CT), in which conventional CT is greater than 20mm or spiral CT is greater than 10mm.
6. Has a life expectancy of at least 3 months.
7. Has a performance status of 0 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
8. Has adequate organ function.
9. Patients with asymptomatic or mild brain metastasis may be enrolled.
10. If female of childbearing potential, is willing to use adequate contraception for the course of the study through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.
11. If male with a female partner(s) of child-bearing potential, must agree to use adequate contraception starting with the first dose of study medication through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.

Exclusion Criteria:

1. Squamous cell carcinoma (including adenosquamous carcinoma);Small cell lung cancer (including small cell cancer and non-small cell mixed lung cancer).

2.ALK(Anaplastic Lymphoma kinase) positive. 3.Imaging (CT or MRI) showed that the tumor lesion invaded the central tumor of local large blood vessels;Or there is obvious pulmonary cavitation or necrotic tumor.

4.History and complications

1. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.(patients with brain metastasis who have completed treatment 14 days before enrollment and have stable symptoms can be included in the group, but they need to be confirmed as having no symptoms of cerebral hemorrhage by brain MRI, CT).
2. Have Participated in other clinical studies or less than 4 weeks before the end of treatment in the previous clinical study.
3. Other active malignancies requiring concurrent treatment.
4. Known history of prior malignancy except if participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy, except for successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
5. Patients who have not recovered to level 1 or lower of NCI-CTCAE4.0 （The Common Terminology Criteria for Adverse Events 4.0）after previous systemic anti-tumor treatment with anti-tumor treatment-related adverse reactions (except hair loss).
6. Abnormal coagulation function (INR(international normalized ratio) >1.5 or PT(prothrombin time) > ULN+4 s or APTT(activated partial thromboplastin time ) > 1.5ULN), with bleeding tendency or receiving thrombolytic or anticoagulant treatment.
7. Is expected to require any other form of antineoplastic therapy while on study.
8. Received a live-virus vaccination within 30 days of planned start of study medication.
9. Known sensitivity to any component of Anlotinib or Sintilimab.
10. Has active autoimmune disease that has required systemic treatment in past 2 years.
11. Is on chronic systemic steroids.
12. Has an active infection requiring therapy.
13. Has known history of Human Immunodeficiency Virus (HIV).
14. Has known active Hepatitis B or C.
15. Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
16. Is a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
17. Has symptomatic ascites or pleural effusion.
18. Has interstitial lung disease or a history of pneumonitis that required oral of IV glucocorticoids to assist with management.
19. Two or more combination therapies for hypertension that are still uncontrollable (systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg).
20. Arteriovenous thrombosis events occurred within 12 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism.
21. clinically significant hemoptysis occurred within 3 months before enrollment (hemoptysis > 50ml daily);Or bleeding symptoms of significant clinical significance or with a clear bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer, baseline stool occult blood ++ or above, or suffering from vasculitis.
22. factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction.
23. Is pregnant or breastfeeding, or expecting to conceive or father children prior to 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  PFS was defined as the time from randomization to documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) or death due to any cause, whichever occurred first and was based on blinded independent central radiologists' (BICR) review. Progressive Disease (PD) was defined as ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. (Note: the appearance of one or more new lesions was also considered progression). Participants were evaluated every 9 weeks with radiographic imaging to assess their response to treatment.

SECONDARY OUTCOMES:
Over Survival(OS) | 2years
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. In those instances where participants were confirmed to be alive on the visit cut-off date of 09 May 2016, survival was censored as of 09 May 2016.
Objective Response Rate (ORR) | 2yeas
  ORR was defined as the percentage of participants in the analysis population who experienced a Complete Response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on BICR evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M.D., Study Chair — The First Hospital of Shijiazhuang
Locations (1):
- The First Hospital of Shijiazhuang, Shijiazhuang, Hebei, China